CLINICAL TRIAL: NCT05637112
Title: ASTER: Anifrolumab Study for Treatment Effectiveness in the Real World Multi-National, Observational, Post-Launch Effectiveness Study Among SLE Patients Receiving Anifrolumab in Routine Clinical Practice
Brief Title: A Treatment Effectiveness Study Among SLE Patients Receiving Anifrolumab in Routine Clinical Practice
Acronym: ASTER
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Other Study IDs: D3461R00043
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: chronic autoimmune disease; immunosuppressants; corticosteroids; human monoclonal antibody (IgG1ƙ mAb); Real World
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prospective Cohort: All patients aged ≥18 years diagnosed with SLE who initiate anifrolumab as prescribed by their healthcare provider (HCP) per the approved country-specific label and are treated at the study sites will be eligible for inclusion.
  Interventions: Other: None (Observational study)

INTERVENTIONS:
Other: None (Observational study) — Not Applicable since Observational Study
  Other Names: Observational Study

SUMMARY:
Anifrolumab Study of Treatment Effectiveness in the Real World (ASTER) study will collect real world data to obtain a good understanding of the (sustained) clinical effect and patient quality of life outcomes among diagnosed SLE patients who initiate anifrolumab treatment. ASTER will generate critical real-world evidence on the benefits of adding anifrolumab to standard of care treatment for SLE in routine clinical practice, to inform physicians, payers and patients.

DETAILED DESCRIPTION:
ASTER is a multi-country, single-arm, prospective, observational study. The study will be initiated on a country-by country basis following the commercial launch of anifrolumab. ASTER is a cohort study, with 1-year retrospective baseline data and 5 years of follow-up data.

The minimum enrolment period is anticipated to be 18 months (± 5 months) per country, but it may be extended, if necessary, to reach the overall study target.

In general, patients will enter the study between the first anifrolumab prescription and infusion (index), with follow-up until death, loss to follow-up, patient discontinuing the study, or end of study period (whichever occurs first). Data collection will continue for all patients including those who have discontinued anifrolumab during the study, unless the patients have withdrawn their consent for participation in the study. Relevant clinical data collection will continue for the entire follow up while patient reported outcome (PRO) data collection will continue only up to the 3-year follow up.

The study will use clinical assessments that are relevant for SLE-treating physicians in routine clinical practice, as well as introduce a specific measure for skin manifestations to affirm the potency of anifrolumab in treating SLE-related skin manifestations.

The eCRFs will be accessed through secure web-based portals and will be used to ensure consistent data collection for each healthcare provider involved in this study.

Electronic data collection will be the only method of data collection in this study.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilled the 2019 EULAR (European League Against Rheumatism)/ACR (American College of Rheumatology) criteria for SLE at the time of study entry.
* Prescribed anifrolumab for their SLE treatment for the first time, according to approved country-specific label.
* The Physician's decision to prescribe anifrolumab must occur prior to any study-related discussion.
* In countries where prescription reimbursements are authorised on a case-by-case basis, authorisation (ie, patient access to treatment) will be required for study entry.

Exclusion Criteria:

* Currently participating in an anifrolumab early access/compassionate use program or an interventional clinical trial with an investigational product.
* Any previous exposure to anifrolumab (including as part of a clinical trial or early access programme).
* Documented diagnosis of severe or rapidly progressive Class III or IV glomerulonephritis requiring induction therapy (mycophenolate mofetil [MMF]/cyclophosphamide [CYC] + high dose steroids), isolated Class V lupus nephritis (in absence of other SLE manifestations, ie. skin/joint involvement), or active severe or unstable neuropsychiatric lupus.
* Any other condition which the investigator deems to limit a patient's ability to understand the informed consent.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged ≥18 years diagnosed with SLE who initiate anifrolumab as prescribed by their healthcare provider (HCP) per the approved country-specific label and are treated at the study sites will be eligible for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 551 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease activity assessed by the Physician Global Assessment (PGA) | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  The PGA is a single-item visual analogue scale that describes the physician assessment of a patient's disease and its impact on daily functioning at the time of assessment. The scale ranges from 0 (asymptomatic disease and no limitation of normal activities) to 3 (severe disease and limitation of normal activities).
Disease activity assessed by Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  The SLEDAI-2K is a global index and includes 24 clinical symptoms and laboratory variables that are weighted by the type of manifestation, but not by severity or dynamic of the individual item. The SLEDAI-2K includes scoring for antibodies and low complement, as well as some renal and hematologic parameters. The total score ranges between 0 and 105, with higher scores representing increased disease activity.
Proportion of patients attaining the composite endpoint of lupus low disease activity (LLDAS) | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  The proportion of patients attaining the composite endpoint of LLDAS will be assesed.

SECONDARY OUTCOMES:
Proportion of patients attaining Definition of Remission in SLE (DORIS) | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  The proportion of patients attaining the Definition of Remission in SLE will be assesed.
Clinical SLE Flares assessment by modified revised Safety of Estrogens in Lupus National Assessment-Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) flare index (rSFI) | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  Flare will be defined as any one criterion present either the Mild/Moderate Flare or Severe Flare categories. New or worsened manifestation will only be reported for manifestation of SLE.
Proportion of patients with irreversible organ damage, using the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SDI). | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  The proportion of patients with irreversible organ damage, using the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index will be assessed. The irreversible, accumulated organ damage from either the disease process or disease treatment, which has been present for at least 6 months, in 12 organ systems will be measured.
SLE treatment patterns prior to, concomitant with and after anifrolumab | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  SLE treatment patterns will be analyzed through prevalence and incidence in respect to time to discontinuation.
Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-Fatigue) | From Baseline (1 year pre-anifrolumab) until follow-up 3 years post-anifrolumab initiation
  The FACIT-Fatigue is a 13-item questionnaire formatted for self-administration that assesses patient-reported fatigue and its impact upon daily activities and function over the past 7 days. Patients will be asked to answer each question using a 5-point verbal rating scale, with total scores ranging from 0 (most fatigued) to 52 (least fatigued).
Lupus Quality of Life (LupusQoL) | From Baseline (1 year pre-anifrolumab) until follow-up 3 years post-anifrolumab initiation
  The LupusQoL is a validated SLE-specific HRQoL (health-related quality of life) instrument consisting of 34 items across 8 domains (Physical health, Emotional health, Body image, Pain, Planning, Fatigue, Intimate relationships, and Burden to others). The LupusQoL has a 5-point verbal rating scale, and uses a 4-week recall period. The mean raw domain score is transformed to scores ranging from 25 (worst HRQoL) to 125 (best HRQoL) by dividing by 4 and then multiplying by 100.
Patient Global Assessment (PtGA) | From Baseline (1 year pre-anifrolumab) until follow-up 3 years post-anifrolumab initiation
  The PtGA is a single-item question that takes into account all the ways in which illness and health conditions may affect the patient at this time. The patient should consider the previous week when answering this question. Responses range from 0 (Very Well) to 100 (Very Poorly) on a visual analogue scale (VAS).
EuroQol 5-Dimension Health Questionnaire 5 Level (EQ-5D-5L) | From Baseline (1 year pre-anifrolumab) until follow-up 3 years post-anifrolumab initiation
  The EQ-5D-5L is a general health status measure comprising a descriptive system and the EQ VAS. The descriptive system comprises 5 dimensions: Mobility, Self-care, Usual activities, Pain/discomfort and Anxiety/depression. Patients are asked to rate their current health and functional status on a 5-point verbal rating scale for each of the 5 domains. Responses are converted into an overall quality of life score via a preference-based statistical mapping algorithm. The scores on these 5 dimensions can be presented as a health profile or can be converted to a single summary index number (utility) reflecting preferability compared to other health profiles. Additionally, patients are asked to indicate how they rate their current overall health on a visual analog scale (EQ-VAS) ranges from 100 for best imaginable health state to 0 for worst imaginable health state.
Work Productivity and Activity Impairment - Lupus (WPAI:lupus) | From Baseline (1 year pre-anifrolumab) until follow-up 3 years post-anifrolumab initiation
  The WPAI:Lupus is an SLE-specific, self-administered questionnaire, that assesses the impact of disease on productivity. The WPAI:Lupus consists of 6 items and has a recall period of the past 7 days. The WPAI:Lupus is divided into 4 domains: Absenteeism (work time missed), Presenteeism (VAS [scored from 0 to 10] rating of impairment while working), Working Productivity Loss (overall work impairment/absenteeism plus presenteeism), and Activity Impairment (VAS [scored from 0 to 10] rating of daily activity, other than work at a job). Scores for each domain are expressed as impairment percentages, with higher scores indicating greater productivity impairment.
Pain Numerical Rating Scale (NRS) | From Baseline (1 year pre-anifrolumab) until follow-up 3 years post-anifrolumab initiation
  The pain NRS will measure the pain severity in the past seven days on a scale of 0-10 (0: no pain; 10: worst pain imaginable).
Number of outpatient hospital and emergency room visits and procedures | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  The healthcare resource utilisation (HCRU) for SLE after anifrolumab initiation as recorded in medical records will be assessed. The number of outpatient hospital and emergency room visits and procedures.
Number of hospital admissions and inpatient hospital procedures | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  The HCRU for SLE after anifrolumab initiation as recorded in medical records will be assessed. The number of hospital admissions and inpatient hospital procedures (including duration of hospital stay and reason for hospitalization, stratified by admission to an intensive care unit [ICU] vs non-ICU) will be assessed.
Number of rheumatologist visits and procedures | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  The HCRU for SLE after anifrolumab initiation as recorded in medical records will be assessed. The number of rheumatologist visits and procedures (including SLE-related laboratory tests) will be assessed.
Number of dialysis appointments | From Baseline (1 year pre-anifrolumab) until follow-up 5 years post-anifrolumab initiation
  The HCRU for SLE after anifrolumab initiation as recorded in medical records will be assessed. The number of dialysis appointments will be assessed.

CONTACTS AND LOCATIONS:
Locations (71):
- Austria (3):
  - Research Site, Innsbruck, Tyrol
  - Research Site, Linz, Upper Austria
  - Research Site, Vienna
- Belgium (4):
  - Research Site, Liège, Li Ge
  - Research Site, Aalst, Oost-Vlaanderen
  - Research Site, Bruges, West Flanders
  - Research Site, Leuven
- Canada (8):
  - Research Site, Calgary, Alberta
  - Research Site, Winnipeg, Manitoba
  - Research Site, Hamilton, Ontario
  - Research Site, Orillia, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Rimouski, Quebec
  - Research Site, Sherbrooke, Quebec
  - Research Site, Ste-Foy, Quebec
- France (14):
  - Research Site, Nice, Alpes-Maritimes
  - Research Site, Clermont-Ferrand, Auvergne-Rh ne-Alpes
  - Research Site, Strasbourg, Bas-Rhin
  - Research Site, Finist Re, Brest Cedex
  - Research Site, Dijon, C te-d'Or
  - Research Site, Bordeaux, Gironde
  - Research Site, Grenoble, Is Re
  - Research Site, Saint-Denis, La R Union
  - Research Site, Nantes, Loire-Atlantique
  - Research Site, Bouches-du-Rh Ne, Lyon
  - Research Site, FORT de France Cedex, Martinique
  - Research Site, Lille, Nord
  - Research Site, Seine-Maritime, Rouen
  - Research Site, Paris
- Germany (14):
  - Research Site, Heidelberg, Baden-W Rttemberg
  - Research Site, Heidelberg, Baden-Wurttemberg
  - Research Site, Erlangen, Bavaria
  - Research Site, Bad Bramstedt, Hamburg
  - Research Site, Schleswig-Holstein, L Beck
  - Research Site, Greifswald, Mecklenburg-Vorpommern
  - Research Site, Munich, Monachium
  - Research Site, Cologne, North Rhine-Westphalia
  - Research Site, D Sseldorf, North Rhine-Westphalia
  - Research Site, Herne, North Rhine-Westphalia
  - Research Site, Mainz A. Rhein, Rhineland-Palatinate
  - Research Site, Magdeburg, Saxony-Anhalt
  - Research Site, Greifwald, Vorpommern-Greifswald
  - Research Site, Berlin
- Israel (8):
  - Research Site, Kfar Saba, Central District
  - Research Site, Tel Hashomer, Central District
  - Research Site, Tiberias, Galilee
  - Research Site, Haifa, Haifa District
  - Research Site, Jerusalem, Jerusalem
  - Research Site, Afula, Northern District
  - Research Site, Ramat Gan, Tel Aviv
  - Research Site, Tel Aviv, Tel Aviv
- Italy (14):
  - Research Site, Napoli, Campania
  - Research Site, Cona, Emilia-Romagna
  - Research Site, Udine, Friuli Venezia Giulia
  - Research Site, Rome, Lazio
  - Research Site, Brescia, Lombardy
  - Research Site, Milan, Lombardy
  - Research Site, Turin, Piedmont
  - Research Site, Cagliari, Sardinia
  - Research Site, Ancona
  - Research Site, Bari
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Pisa
  - Research Site, Roma
- Sweden (3):
  - Research Site, Örebro, N Rke
  - Research Site, Danderyd, Stockholm County
  - Research Site, Stockholm, Uppland
- United Arab Emirates (3):
  - Research Site, Dubai, Dubayy
  - Research Site, Sharjah city, Emirate of Sharjah
  - Research Site, Abu Dhabi

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Mosca M, Emmas C, Nekeman-Nan C, Stirnadel-Farrant H, Chen S, Carty L, Waratani M, Seo C, Chen S, Sorrentino A. Anifrolumab Study for Treatment Effectiveness in the Real World (ASTER) among patients with systemic lupus erythematosus: protocol for an international observational effectiveness study. BMJ Open. 2024 Nov 21;14(11):e086055. doi: 10.1136/bmjopen-2024-086055. PMID 39578022